CLINICAL TRIAL: NCT06845202
Title: A Phase 1/2, Randomized, Double-blind, Placebo-controlled 2-part Study of the Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of Single Dose ALN-4324 in Overweight to Obese Adult Healthy Volunteers and Multiple Dose ALN-4324 in Overweight to Obese Patients With Type 2 Diabetes Mellitus (T2DM)
Brief Title: A Study to Evaluate ALN-4324 in Overweight to Obese Healthy Volunteers and in Overweight to Obese Patients With T2DM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALN-4324-001; 2024-519005-35-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Obese or Overweight Healthy Volunteers; Type 2 Diabetes Mellitus (T2DM)
Keywords: siRNA; RNAi therepeutic
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: ALN-4324 (Experimental): Participants will be administered a single dose of ALN-4324.
  Interventions: Drug: ALN-4324
- Part A: Placebo (Placebo Comparator): Participants will be administered a single dose of placebo.
  Interventions: Drug: Placebo
- Part B: ALN-4324 (Experimental): Participants will be administered multiple doses of ALN-4324
  Interventions: Drug: ALN-4324
- Part B: Placebo (Placebo Comparator): Participants will be administered multiple doses of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALN-4324 — ALN-4324 will be administered subcutaneously (SC)
  Arms: Part A: ALN-4324; Part B: ALN-4324
Drug: Placebo — Placebo will be administered SC
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The purpose of this study is to:

* evaluate the safety and tolerability of single ascending doses of ALN-4324 in healthy volunteers and to characterize the single-dose PK of ALN-4324
* evaluate the efficacy, safety, tolerability, and pharmacodynamics (PD) of multiple doses of ALN-4324 in adult overweight to obese patients with T2DM

ELIGIBILITY:
Inclusion Criteria:

Part A:

* Has a body mass index (BMI) of ≥27 kg/m^2 and <40 kg/m^2

Part B:

* Is an adult patient with a confirmed diagnosis of T2DM
* Has a hemoglobin A1c (HbA1c) ≥7% to <10.5%
* Has a BMI of ≥25 kg/m^2 and <45 kg/m^2
* Is on a stable dose of either metformin or metformin and a sodium-glucose cotransporter 2 inhibitor (SGLT2i)

Exclusion Criteria:

Part A:

* Has known human immunodeficiency virus (HIV) infection; or known current or chronic hepatitis C virus or hepatitis B virus infection

Part B:

* Receiving therapies for chronic weight management or antidiabetic medications other than metformin and SGLT2i

Note: other protocol defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Part A: Frequency of Adverse Events (AEs) | Up to 9 months
Part B: Frequency of Adverse Events | Up to 12 months

SECONDARY OUTCOMES:
Part A: Area Under the Plasma Concentration-time Curve (AUC) of ALN-4324 in Plasma | Predose and up to 3 days postdose
Part A: Maximum Observed Plasma Concentration (Cmax) of ALN-4324 in Plasma | Predose and up to 3 days postdose
Part A: Time to Maximum Plasma Concentration (Tmax) of ALN-4324 in Plasma | Predose and up to 3 days postdose
Part A: Fraction of ALN-4324 excreted in urine | Predose and up to 24 hours postdose (fe)
Part B: Change from Baseline in HbA1c | Baseline up to 6 months
Part B: Response to Glucose Tolerance Test | Predose and up to 2 hours postdose
Part B: Concentrations of ALN-4324 in Plasma | Predose and up to 4 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (20):
- United States (7):
  - Clinical Trial Site, Montclair, California
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, Overland Park, Kansas
  - Clinical Trial Site, Berlin, New Jersey
  - Clinical Trial Site, Monroe, North Carolina
  - Clinical Trial Site, Raleigh, North Carolina
- Argentina (3):
  - Clinical Trial Site, Mar del Plata, B
  - Clinical Trial Site, San Miguel de Tucumán, T
  - Clinical Trial Site, Buenos Aires
- Canada (3):
  - Clinical Trial Site, Vancouver, British Columbia
  - Clinical Trial Site, Concord, Ontario
  - Clinical Trial Site, Mount Royal, Quebec
- Clinical Trial Site, Santiago, RM, Chile
- Germany (2):
  - Clinical Trial Site, Essen, Northwest
  - Clinical Trial Site, Essen
- Poland (4):
  - Clinical Trial Site, Gdansk
  - Clinical Trial Site, Lublin
  - Clinical Trial Site, Tarnów
  - Clinical Trial Site, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Access to data may be declined where there is likelihood a patient could be identified or other feasibility issue, where there is a potential conflict of interest, planned business activities or an actual or potential competitive risk. Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Timeframes for data access may vary and can take up to 6 months or more.
  Requests for access to data can be submitted via the website www.vivli.org. Questions can also be directed to datasharing@alnylam.com.